CLINICAL TRIAL: NCT03720067
Title: Propranolol, Carvedilol and Rosuvastatin in the Prevention of Recurrent Variceal Haemorrhage in Patients With Cirrhotic Portal Hypertension
Brief Title: Propranolol, Carvedilol and Rosuvastatin in the Prevention of Variceal Bleeding in Cirrhotic Portal Hypertension
Acronym: Betastatin
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Guilherme Rezende, Associated Professor, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 83211318.1.0000.5257
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Cirrhosis; Portal Hypertension; Variceal Hemorrhage
MeSH Terms: conditions — Fibrosis; Hypertension, Portal | interventions — Propranolol; Carvedilol; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Phase 1: Propranolol (PPL) (Active Comparator): Hepatic venous pressure gradient (HVPG) will be measured before and after 120 minutes of a loading dose of Propranolol (PPL) 80 mg PO. Thereafter, patients will receive maintenance therapy with Propranolol (40 to 320 mg / day) adjusted according to blood pressure and heart rate. After 28 days of reaching the maximum tolerated dose, a new HVPG measurement will be performed.
  Interventions: Drug: Propranolol
- Phase 1: Carvedilol (CVD) (Active Comparator): HVPG will be measured before and after 120 minutes of a loading dose of Carvedilol (CVD) 12.5 mg PO. Thereafter, patients will receive maintenance therapy with Carvedilol (6.25 - 25 mg / day) adjusted according to blood pressure. After 28 days of reaching the maximum tolerated dose, a new HVPG measurement will be performed.
  Interventions: Drug: Carvedilol
- Phase 2: PPL non-responders/rosuvastatin (Active Comparator): Patients treated with PROPRANOLOL (PPL) who do not reach HVPG fall below 12 mmHg will be randomized to receive the addition of ROSUVASTATIN 20 mg /day PO. HVPG will be measured again after 56 days.
  Interventions: Drug: Propranolol; Drug: Rosuvastatin
- Phase 2: PPL non-responders/placebo (Placebo Comparator): Patients treated with PROPRANOLOL (PPL) who do not reach HVPG fall below 12 mmHg will be randomized to receive the addition of PLACEBO 1 tablet PO. HVPG will be measured again after 56 days.
  Interventions: Drug: Propranolol; Drug: Placebo
- Phase 2: CVD non-responders/rosuvastatin (Active Comparator): Patients treated with CARVEDILOL (CVD) who do not reach HVPG fall below 12 mmHg will be randomized to receive the addition of ROSUVASTATIN 20 mg /day PO. HVPG will be measured again after 56 days.
  Interventions: Drug: Carvedilol; Drug: Rosuvastatin
- Phase 2: CVD non-responders/placebo (Placebo Comparator): Patients treated with CARVEDILOL (CVD) who do not reach HVPG fall below 12 mmHg will be randomized to receive the addition of PLACEBO 1 tablet PO. HVPG will be measured again after 56 days.
  Interventions: Drug: Carvedilol; Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — 40mg to 320mg / day
  Arms: Phase 1: Propranolol (PPL); Phase 2: PPL non-responders/placebo; Phase 2: PPL non-responders/rosuvastatin
Drug: Carvedilol — 6.25mg to 25mg / day
  Arms: Phase 1: Carvedilol (CVD); Phase 2: CVD non-responders/placebo; Phase 2: CVD non-responders/rosuvastatin
Drug: Rosuvastatin — 20mg / day
  Arms: Phase 2: CVD non-responders/rosuvastatin; Phase 2: PPL non-responders/rosuvastatin
Drug: Placebo — Placebo of rosuvastatin
  Arms: Phase 2: CVD non-responders/placebo; Phase 2: PPL non-responders/placebo

SUMMARY:
Patients with hepatic cirrhosis and previous variceal bleeding will be randomly assigned to use propranolol or carvedilol. After 8 weeks, rosuvastatin or placebo will be blindly added to nonresponders (HVPG measurement > 12mmHg) for another 8 weeks and hemodynamic response will be assessed again.

Surrogate serum markers of portal hypertension will be evaluated and correlated to HVPG values and to its variations.

ELIGIBILITY:
Inclusion Criteria:

* Hepatic cirrhosis of any etiology
* Previous variceal bleeding
* Endoscopic variceal eradication at least 2 weeks before

Exclusion Criteria:

* Beta blocker or statin contraindications
* Model for End-Stage Liver Disease (MELD) score > 25
* Child-Pugh score > 13
* HVPG ≤ 12 mmHg
* Creatinine clearance < 50 mL/min
* Refractory ascites
* Hepatic encephalopathy stages 3 or 4
* Alcohol use in the last 6 months
* Hepatitis C treatment in the last 6 months
* Changing or initiating a new hepatitis B treatment in the last 6 months
* Malignant neoplasms from any origin except basal cell carcinoma
* HIV infection
* Pregnancy
* Anticoagulation
* Recent or complete portal vein thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-01-25 (Actual); Primary Completion 2020-12-20 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Acute hemodynamic response | Two hours after a load dose of carvedilol or propranolol
  A decrease in HVPG to 12 mmHg or lower
Full hemodynamic response to beta blockers | Eight weeks of carvedilol or propranolol
  A decrease in HVPG to 12 mmHg or lower
Full hemodynamic response to beta blockers plus rosuvastatin or placebo | Eight weeks of beta blockers plus rosuvastatin or placebo
  A decrease in HVPG to 12 mmHg or lower

SECONDARY OUTCOMES:
Sufficient hemodynamic response to beta blockers plus rosuvastatin or placebo | Eight weeks of beta blockers plus rosuvastatin or placebo
  A decrease in HVPG of at least 20% from baseline
Partial hemodynamic response to beta blockers plus rosuvastatin or placebo | Eight weeks of beta blockers plus rosuvastatin or placebo
  A decrease in HVPG of at least 10% from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal do Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No